CLINICAL TRIAL: NCT04928534
Title: Observational Cohort Study of Blood Transcriptomics and Proteomics Information as Biomarkers of Traumatic Encephalopathy Syndrome
Brief Title: Cohort Study of Blood Biomarkers for TES
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Xintong Ge, Principal Investigator, Tianjin Medical University General Hospital
Other Study IDs: IRB2021-YX-056-01
Record Dates: First submitted 2021-06-06; First posted 2021-06-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Traumatic Encephalopathy; Traumatic Encephalopathy, Chronic; Traumatic; Encephalopathy, Postcontusional
MeSH Terms: conditions — Chronic Traumatic Encephalopathy; Brain Diseases | interventions — Hematologic Tests; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Athletes with rmTBI history: 50 active or retired athletes from the Weightlifting, Wrestling, Judo, Boxing and Taekwondo Sports Management Center of Tianjin Sports Bureau
  Interventions: Diagnostic Test: Blood tests, Cognitive function tests, head MRI (plain scan and DTI sequence) examination and head PET (FDG-PET, Tau-PET and Amyloid-PET) examination
- Patients with rmTBI history: 50 patients with multiple (≥2 times) exposure to brain trauma attending Tianjin Medical Insurance designated hospitals such as Tianjin Medical University General Hospital
  Interventions: Diagnostic Test: Blood tests, Cognitive function tests, head MRI (plain scan and DTI sequence) examination and head PET (FDG-PET, Tau-PET and Amyloid-PET) examination
- Healthy volunteer: 20 healthy volunteers
  Interventions: Diagnostic Test: Blood tests, Cognitive function tests, head MRI (plain scan and DTI sequence) examination and head PET (FDG-PET, Tau-PET and Amyloid-PET) examination

INTERVENTIONS:
Diagnostic Test: Blood tests, Cognitive function tests, head MRI (plain scan and DTI sequence) examination and head PET (FDG-PET, Tau-PET and Amyloid-PET) examination — 1. Blood tests (30-ml venous blood) for the following items. 1) Transcriptomics and proteomics high-throughput detection and quantitative verification; 2) Exosomal transcriptomics and proteomics high-throughput detection and quantitative verification; 3) Quantitative detection for classical biomarkers of traumatic brain injury, including S100B, GFAP, UCH-L1, NFL, T-Tau and p-Tau181.
  2. Cognitive function tests, including RPQ, MMSE and MoCA.
  3. Possible head MRI (plain scan and DTI sequence) examination and head PET (FDG-PET, Tau-PET and Amyloid-PET) examination

SUMMARY:
In this study, high-throughput screening and multi-omics (transcriptomics and proteomics) joint analysis technology will be employed to explore potential CTE/TES biomarkers (RNA and protein) in blood and its exosomes. Thereafter, these biomarkers will be combined with the reported TBI biomarkers to create a novel set of CTE/TES molecular diagnostic signatures. The findings may open a new avenue for the clinical diagnosis of the disease and the future research on its therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Athletes and patients with traumatic brain injury

   * Age ≥ 18 and ≤ 80 years old with independent behavior ability or authorized legal representative.
   * Have a clear history of repetitive mild TBI, concussion or subconcussion.
   * The most recent head injury occurred 3 months ago.
2. Healthy Volunteers

   * Age ≥ 18 and ≤ 80 years old with independent behavior ability.
   * No history of repetitive mild TBI, concussion or subconcussion.
   * Fully understands the nature of the study, and voluntarily participates and signs the informed consent.

Exclusion Criteria:

1. Athletes and patients with traumatic brain injury

   * Pregnant or lactating women.
   * History of other neurological diseases.
   * History of tumors, hematological diseases, severe cardiopulmonary diseases, hepatic failure or renal failure.
   * Have participated in clinical trials in the past four weeks.
   * The investigator believes that not appropriate for inclusion.
2. Healthy Volunteers

   * Pregnant or lactating women.
   * History of TBI or other neurological diseases.
   * History of tumors, hematological diseases, severe cardiopulmonary diseases, hepatic failure or renal failure.
   * Have participated in clinical trials in the past four weeks.
   * The investigator believe that not appropriate for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Athletes with rmTBI history. The subjects are active or retired athletes who have engaged in weightlifting, wrestling, judo, boxing or taekwondo. All of them have a clear history of rmTBI.
  * Patients with rmTBI history. The subjects have a history of multiple (≥2 times) exposure to brain trauma, and medical records in Tianjin Medical Insurance designated hospitals.
  * Healthy volunteers, without rmTBI history.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Blood level of novel protein biomarkers for CTE/TES | Baseline
  Novel protein biomarkers for CTE/TES will be screened out by transcriptomics + proteomics high-throughput detection and multi-omics bioinformatics analysis. Their levels will be further verified using ELISA assay.
Blood level of novel RNA biomarkers for CTE/TES | Baseline
  Novel RNA biomarkers for CTE/TES will be screened out by transcriptomics + proteomics high-throughput detection and multi-omics bioinformatics analysis. Their levels will be further verified using RT-PCR.

SECONDARY OUTCOMES:
Blood level of classical biomarkers for CTE/TES | Baseline
  Blood S100B, GFAP, UCH-L1, NFL, T-Tau and p-Tau181 level detected by ELISA assay
Ultrasound examination of the carotid arteries and lower limb arteries | 5 years post-enrollment
  Ultrasound examination of bilateral CCA, ICA, CFA, SFA, PA, DPA and ATA
Serum Treg cell count and degree of senescence | 5 years post-enrollment
  Percentage of serum regulatory T (Treg) cells relative to the total T cell count; Percentage of senescent Treg cells relative to the total Treg cell count
Cognitive function tests - RPQ-3 | 5 years post-enrollment
  Rivermead post-concussion symptoms questionnaire - 3 (RPQ-3). Reference Range: 0-12. Higher scores mean a worse outcome.
Cognitive function tests - RPQ-16 | 5 years post-enrollment
  Rivermead post-concussion symptoms questionnaire - 16 (RPQ-16). Reference Range: 0-64. Higher scores mean a worse outcome.
Cognitive function tests - MoCA | 5 years post-enrollment
  Montreal cognitive assessment (MoCA). Reference Range: 0-30. Higher scores mean a better outcome.
Cognitive function tests - MMSE | 5 years post-enrollment
  Description: mini-mental state examination (MMSE). Reference Range: 0-30. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lei, Doctor, Principal Investigator — Tianjin Medical University
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04928534/Prot_000.pdf
  • Informed Consent Form (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04928534/ICF_001.pdf